CLINICAL TRIAL: NCT00596726
Title: RECOVER I: IMPELLA® RECOVER® LP/LD 5.0 Support System: A Clinical Safety & Feasibility Study
Brief Title: RECOVER I Impella RECOVER LP/LD 5.0 Support System Safety and Feasibility Study
Acronym: RECOVER I
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abiomed Inc. (Industry)
Responsible Party: Bartley Griffith M.D., University of Maryland, MD
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G030202
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2010-05

CONDITIONS: Cardiac Surgery
Keywords: All patients presenting for high-risk cardiac surgery and who might post-operatively meet the study inclusion criteria are potential study candidates.

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: IMPELLA LP/LD 5.0 — IMPELLA LP/LD 5.0 Support System is intended to be used for up to seven (7) days as a left ventricular cardiac assist device for postcardiotomy patients who, despite having been weaned from cardiopulmonary bypass (CPB), require hemodynamic support

SUMMARY:
To demonstrate that that the device is safe and potentially efficacious for use as a left ventricular cardiac assist device for postcardiotomy patients who require hemodynamic support post weaning from cardiopulmonary bypass.

DETAILED DESCRIPTION:
To demonstrate that the device is safe and potentially efficacious for use as a left ventricular cardiac assist device for postcardiotomy patients who require hemodynamic support post weaning from cardiopulmonary bypass. Postcardiotomy patients, weaned from a cardiopulmonary bypass system (CPB) in need for hemodynamic support due to ineffective standard medical therapy will be considered for enrollment. An attempt shall be made to reverse the hemodynamic situation with medications (e.g. inotropes, vasopressors). The IMPELLA RECOVER LP/LD 5.0 will be implanted by the surgeon when no improvement in hemodynamics is observed.

ELIGIBILITY:
Inclusion Criteria:

* BSA
* Receiving stable infusion of one high dose inotrope or two medium dose inotropes for a respective minimum time indicated.
* C.I.
* Elevated Filling Pressures, PCWP or PA
* Time to enrollment within 48 hours from weaning

Exclusion Criteria:

* Renal dysfunction
* Hepatic dysfunction
* Right Ventricular failure defined.
* LV or RV Thrombus
* Other exclusions per protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2006-08; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Frequency of Major Adverse Events | 30 day or discharge

SECONDARY OUTCOMES:
Other Adverse Events Doppler echocardiography assessment of aortic valve function will be performed at explant and 30days and 3 month follow-ups. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Bartley Griffith, M.D., Principal Investigator — University of Maryland; Mark Anderson, Principal Investigator — Robert Wood Johnson Foundation
Locations (7):
- United States (7):
  - University of Maryland, Baltimore, Maryland
  - Massach General Hospital, Boston, Massachusetts
  - Brigham & Womens, Boston, Massachusetts
  - Robert Wood Johnson, New Brunswick, New Jersey
  - Columbia Presbyterian Hospital, New York, New York
  - Hershey Medical Center, Hershey, Pennsylvania
  - Texas Heart, Houston, Texas